CLINICAL TRIAL: NCT03047447
Title: Induced and Controlled Dietary Ketosis as a Regulator of Obesity and Metabolic Syndrome Pathologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristlecone Behavioral Health, Inc. (Industry)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bristlecone Health
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Metabolic Syndrome; Diabetes Mellitus, Type 2; Pre Diabetes
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketogenic group (Experimental): 10-week diet with controlled glycemic indices provided for ketogenic group. Baseline triglyceride, HgA1c, VO2 max, body mass index (BMI), resting metabolic rate (RMR), blood ketone levels and body fat mass measurements were assessed at week 0 and week 3, 6 and 10.
  Interventions: Behavioral: Dietary Ketosis: Regulator of Obesity and Metabolic Syndrome
- Exercise group (Active Comparator): Exercise group maintained normal diet for 10-weeks and exercised 3-5 days per week. Baseline triglyceride, HgA1c, VO2 max, body mass index (BMI), resting metabolic rate (RMR), blood ketone levels and body fat mass measurements were assessed at week 0 and week 3, 6 and 10.
  Interventions: Behavioral: Dietary Ketosis: Regulator of Obesity and Metabolic Syndrome
- Non-exercise (Active Comparator): Non-exercise group maintained normal diet for 10-weeks with no exercise. Baseline triglyceride, HgA1c, VO2 max, body mass index (BMI), resting metabolic rate (RMR), blood ketone levels and body fat mass measurements were assessed at week 0 and week 3, 6 and 10.
  Interventions: Behavioral: Dietary Ketosis: Regulator of Obesity and Metabolic Syndrome

INTERVENTIONS:
Behavioral: Dietary Ketosis: Regulator of Obesity and Metabolic Syndrome — 30 adults previously diagnosed with MetS randomly prescribed to one of three groups: a sustained ketogenic diet with no exercise, the participant's normal diet with no exercise, or participant's normal diet with 3-5 days per week of exercise for 30 minutes

SUMMARY:
Original research article entitled Induced and Controlled Dietary Ketosis as a Regulator of Obesity and Metabolic Syndrome by Madeline Gibas for consideration for publication in a clinical journal. This research manuscript builds on previous landmark studies that report that major weight and fat mass loss in type II (T2D) patients who were fed a very low carbohydrate, ketogenic diet. In this manuscript, the investigators outline our research study that showed statistically significant (p < 0.05) changes over time in hemoglobin A1c, weight, BMI, body fat percentage and ketones for patients with metabolic syndrome who were fed a very low carbohydrate diet, ketogenic diet.

DETAILED DESCRIPTION:
Purpose -Assessment of prolonged, physiological, dietary ketosis on pathological processes induced by metabolic syndrome (MetS) including a reduction in fasting triglycerides, BMI and body fat mass, a significant decrease and/or normalization of HgA1c and an increase in resting metabolic rate.

Design - Qualitative

Setting - Bristlecone Health, Inc., Maple Grove, Minnesota

Subjects - 30 adults previously diagnosed with MetS randomly prescribed to one of three groups: a sustained ketogenic diet with no exercise, the participant's normal diet with no exercise, or participant's normal diet with 3-5 days per week of exercise for 30 minutes.

Intervention - 10-week diet with controlled glycemic indices provided for ketogenic group; other groups maintained normal diet. Baseline triglyceride, HgA1c, VO2 max, body mass index (BMI), resting metabolic rate (RMR), blood ketone levels and body fat mass measurements were assessed for all three groups at week 0 and week 3, 6 and 10.

Measures - ANOVA followed by tests pairwise differences using Tukey's HSD correction.

Analysis - Five of the seven variables for the ketogenic group showed a statistically significant difference between week 0 and 10 data points.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with metabolic syndrome

Exclusion Criteria:

* No diagnosis of metabolic syndrome
* < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bristlecone Behavioral Health, Inc., Maple Grove, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketogenic Group | Exercise Group | Non-exercise
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketogenic Group | Exercise Group | Non-exercise | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Age] | 47.70 (9.51) | 48.20 (9.77) | 50.20 (6.75) | 48.70 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 10 | 26
  Male | 4 | 0 | 0 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c
Description: Hemoglobin A1c (HgA1c) was measured at week 0 and week 3, 6 and 10 for the experimental ketogenic group, the control standard American diet group with no exercise, and the control standard American diet group with 3-5 days of exercise per week (120-150 minutes/week). The change over time was calculated for HgA1c at week 10 minus the HgA1c value at week 0.
Time Frame: Week 0 - Week 10
Measure: Mean (95% Confidence Interval); unit: % of hemoglobin
Groups:
- Ketogenic Group: 10-week diet with controlled glycemic indices provided for ketogenic group. Baseline triglyceride, HgA1c, VO2 max, body mass index (BMI), resting metabolic rate (RMR), blood ketone levels and body fat mass measurements were assessed at week 0 and week 3, 6 and 10.
  Dietary Ketosis: Regulator of Obesity and Metabolic Syndrome: 30 adults previously diagnosed with MetS randomly prescribed to one of three groups: a sustained ketogenic diet with no exercise, the participant's normal diet with no exercise, or participant's normal diet with 3-5 days per week of exercise for 30 minutes.
  p=0.00
- Exercise Group: Exercise group maintained normal diet for 10-weeks and exercised 3-5 days per week. Baseline triglyceride, HgA1c, VO2 max, body mass index (BMI), resting metabolic rate (RMR), blood ketone levels and body fat mass measurements were assessed at week 0 and week 3, 6 and 10.
  Dietary Ketosis: Regulator of Obesity and Metabolic Syndrome: 30 adults previously diagnosed with MetS randomly prescribed to one of three groups: a sustained ketogenic diet with no exercise, the participant's normal diet with no exercise, or participant's normal diet with 3-5 days per week of exercise for 30 minutes.
  p=0.11
- Non-exercise: Non-exercise group maintained normal diet for 10-weeks with no exercise. Baseline triglyceride, HgA1c, VO2 max, body mass index (BMI), resting metabolic rate (RMR), blood ketone levels and body fat mass measurements were assessed at week 0 and week 3, 6 and 10.
  Dietary Ketosis: Regulator of Obesity and Metabolic Syndrome: 30 adults previously diagnosed with MetS randomly prescribed to one of three groups: a sustained ketogenic diet with no exercise, the participant's normal diet with no exercise, or participant's normal diet with 3-5 days per week of exercise for 30 minutes.
  p=.211
Arm/Group | Ketogenic Group | Exercise Group | Non-exercise
Number analyzed (Participants) | 10 | 10 | 10
% of hemoglobin | -.42 [-0.95 to 0.11] | -0.37 [-0.74 to 0.00] | 0.02 [-0.35 to 0.39]
Statistical Analysis 1: Comparison: Ketogenic Group vs Exercise Group vs Non-exercise; Test type: Other; p = 0.001, ANOVA — Change over time from week 0 to week 10 with HgA1c for experimental ketogenic group vs.control exercise and non-exercise groups

2. Secondary Outcome: Weight
Description: Weight was measured at week 0 and week 3, 6 and 10 for the experimental ketogenic group, the control standard American diet group with no exercise, and the control standard American diet group with 3-5 days of exercise per week (120-150 minutes/week). The change over time was calculated for weight at week 10 minus weight at week 0.
Time Frame: 10-weeks
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | Ketogenic Group | Exercise Group | Non-exercise
Number analyzed (Participants) | 10 | 10 | 10
pounds | -28.40 [-34.14 to -23.06] | -2.87 [-7.06 to 0.78] | -2.43 [-6.34 to 1.48]
Statistical Analysis 1: Comparison: Ketogenic Group vs Exercise Group vs Non-exercise; Test type: Other; p = 0.001, ANOVA; Change over time from week 0 to week 10 with weight for experimental ketogenic group vs.control exercise and non-exercise groups

3. Secondary Outcome: BMI (Body Mass Index)
Description: BMI (body mass index) was measured at week 0 and week 3, 6 and 10 for the experimental ketogenic group, the control standard American diet group with no exercise, and the control standard American diet group with 3-5 days of exercise per week (120-150 minutes/week). The change over time was calculated for BMI at week 10 minus BMI at week 0.
Time Frame: 10-weeks
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Ketogenic Group | Exercise Group | Non-exercise
Number analyzed (Participants) | 10 | 10 | 10
kg/m^2 | -4.4 [-5.5 to -3.2] | -0.01 [-0.83 to 0.81] | -0.42 [-1.24 to 0.40]
Statistical Analysis 1: Comparison: Ketogenic Group vs Exercise Group vs Non-exercise; Test type: Other; p = 0.001, ANOVA; Change over time from week 0 to week 10 with BMI for experimental ketogenic group vs.control exercise and non-exercise groups

4. Secondary Outcome: Body Fat Mass (Pounds of Body Fat)
Description: BFM (body fat mass) was measured at week 0 and week 3, 6 and 10 for the experimental ketogenic group, the control standard American diet group with no exercise, and the control standard American diet with 3-5 days of exercise per week (120-150 minutes/week). The change over time was calculated for BFM at week 10 minus BFM at week 0.
Time Frame: 10-weeks
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | Ketogenic Group | Exercise Group | Non-exercise
Number analyzed (Participants) | 10 | 10 | 10
pounds | -0.03 [-0.04 to -0.02] | -0.01 [-0.01 to 0.00] | -0.00 [-0.01 to 0.00]
Statistical Analysis 1: Comparison: Ketogenic Group vs Exercise Group vs Non-exercise; Test type: Other; p = 0.001, ANOVA; Change over time from week 0 to week 10 with body fat mass for experimental ketogenic group vs.control exercise and non-exercise groups

5. Secondary Outcome: Ketones (Blood)
Description: Ketones (blood) were measured at week 0 and week 3, 6 and 10 for the experimental ketogenic group, the control standard American diet group with no exercise, and the control standard American diet with 3-5 days of exercise per week (120-150 minutes/week). The change over time was calculated for ketones (blood) at week 10 minus ketones (blood) at week 0.
Time Frame: 10-weeks
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Ketogenic Group | Exercise Group | Non-exercise
Number analyzed (Participants) | 10 | 10 | 10
mmol/L | 0.24 [0.14 to 0.34] | 0.07 [-0.00 to 0.14] | 0.04 [-0.03 to 0.11]
Statistical Analysis 1: Comparison: Ketogenic Group vs Exercise Group vs Non-exercise; Test type: Other; p = 0.001, ANOVA; Change over time from week 0 to week 10 with blood ketones for experimental ketogenic group vs.control exercise and non-exercise groups

ADVERSE EVENTS:
Arm/Group | Ketogenic Group | Exercise Group | Non-exercise
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No